CLINICAL TRIAL: NCT02916953
Title: Clinical Evaluation of the Safety of a Local Osteo-Enhancement Procedure (LOEP™) Intended to Increase Bone Strength in the Proximal Femur of Women in Europe With Osteoporosis
Brief Title: CONFIRM - Study of AGN1 LOEP in Patients With Osteoporosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AgNovos Healthcare, LLC (Industry)
Collaborators: KCR S.A. (Unknown); genae Group (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRE-EU-101.1
Record Dates: First submitted 2016-09-26; First posted 2016-09-28 (Estimated); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Treatment (Experimental): All subjects who meet the inclusion and exclusion criteria will receive the AGN1 Femoral Local Osteo-Enhancement Procedure (LOEP™) treatment
  Interventions: Device: AGN1 Femoral Local Osteo-Enhancement Procedure

INTERVENTIONS:
Device: AGN1 Femoral Local Osteo-Enhancement Procedure — A procedure that is intended to increase the strength of the proximal femur in individuals with osteoporosis of the femoral neck. Local treatment of the proximal femur with AGN1 is intended to be adjunctive to appropriate systemic therapy and overall osteoporosis management as directed by the patient's treating physicians.
  Other Names: AGN1 Femoral LOEP™

SUMMARY:
The study will evaluate the immediate procedure and post-procedure profile of the AGN1 Femoral LOEP™ Kit. All subjects will receive the treatment and be evaluated for any adverse or serious adverse events that could occur during the procedure or immediately post-procedure.

DETAILED DESCRIPTION:
This research study will be conducted as a post-CE Mark prospective multi-center study within Europe. In total 60 patients will be treated with the OSSURE LOEP kit.

Follow-up visits will be conducted ten (10) and forty-two (42) days after the procedure. In addition, all subjects will have the option to consent for a long term follow-up evaluation at twelve (12) months post-procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is postmenopausal female (at least 1-year post menses).
2. Subject has osteoporosis as defined by a documented DXA scan T score of ≤ -2.5 in the femoral neck of at least one hip within the last year. If no documented T-score, then a DXA scan will be performed during eligibility screening.
3. Subject has one hip without previous surgery or fracture.
4. Subject is medically stable from any previous treatment or medical procedure in the opinion of the investigator and with an ASA score of I or II.
5. Subject has willingness, ability, and commitment to participate in baseline and follow-up evaluations for the full length of the study.
6. Subject is capable of giving written informed consent to participate in the study.

Exclusion Criteria:

1. Subject is less than six (6) months removed from having a hip fracture repair or prosthesis, or less than three (3) months removed from an elective THA.
2. Subject has progressive increase in undiagnosed hip pain over the previous six months that in the opinion of the Investigator may suggest other underlying bone or joint pathology (e.g. rheumatoid arthritis, fracture, etc.).
3. Subject is dependent on the use of a wheel-chair or is bed-ridden.
4. Subject has albumin corrected serum calcium levels outside the normal lab range or has a pre-existing calcium metabolism disorder (e.g. hypercalcemia).
5. Subject has severe renal insufficiency defined as an estimated glomerular filtration rate (eGFR) ≤ 30 mL/min or is being treated with dialysis.
6. Subject has insulin-dependent diabetes mellitus (IDDM).
7. Subject has Body Mass Index (BMI) > 35.
8. Subject exhibits excessive smokeless tobacco use or excessive smoking as determined by the principal investigator*.
9. Subject exhibits excessive alcohol consumption as determined by the principal investigator*.
10. Subject has radiological evidence of gross bony or joint pathology, including signs predictive of atypical femoral fractures (e.g. Cortical beaking) or has been diagnosed and/or treated for atypical femoral fractures.
11. Subject treated with corticosteroids or systemic glucocorticoids for ten (10) days in the previous six (6) months.
12. Subject has history of oral or parenteral use of immune-suppressive drugs in the previous twelve months.
13. Subject has history of metabolic bone disease other than osteoporosis (ex. Paget's disease).
14. Subject has a history of auto-immune arthritic diseases including rheumatoid, psoriatic, or those associated with systemic lupus erythematosus, spondyloarthropathy, Reiter's Syndrome or Crohn's Disease.
15. Subject has a history of radiation therapy to the hip or pelvic region.
16. Subject has a history of any invasive malignancy (except basal cell carcinoma), unless treated and with no clinical signs of symptoms of malignancy for five (5) years.
17. Subject has known allergies to implanted device.
18. Subject has severe comorbidity or poor general physical/mental health that, in the opinion of the Investigator, will not allow the subject to be a good study candidate.
19. Subject is currently enrolled in another clinical study. *AgNovos's recommendation is >1 pack per day smoking and >3 alcoholic drinks per day

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-12-17 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2022-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with procedure-related or device-related adverse events | 42 Days
  Adverse Events and Serious Adverse Events related to either the treatment or device.
  The incidence of all adverse events occurring during the first forty-two (42) day follow-up period determined to be at least possibly related to the procedure and/or device for the local treatment of osteoporosis.

CONTACTS AND LOCATIONS:
Overall Officials: Jo De Schepper, MD, Principal Investigator — AZ Nikolaas
Locations (5):
- Belgium (4):
  - AZ Sint-Blasius, Dendermonde
  - AZ Maria Middelares, Ghent
  - AZ Groeninge - Campus Kennedylaan, Kortrijk
  - AZ Sint-Nikolaas, Sint-Niklaas
- Maastricht UMC, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Decision on what data to share has not yet been determined.

REFERENCES:
- [Background] International Osteoporosis Foundation. Facts and Statistics. 2013: http://www.iofbonehealth.org/facts-statistics.
- [Background] MacLean C, Newberry S, Maglione M, McMahon M, Ranganath V, Suttorp M, Mojica W, Timmer M, Alexander A, McNamara M, Desai SB, Zhou A, Chen S, Carter J, Tringale C, Valentine D, Johnsen B, Grossman J. Systematic review: comparative effectiveness of treatments to prevent fractures in men and women with low bone density or osteoporosis. Ann Intern Med. 2008 Feb 5;148(3):197-213. doi: 10.7326/0003-4819-148-3-200802050-00198. Epub 2007 Dec 17. PMID 18087050
- [Background] Abrahamsen B, van Staa T, Ariely R, Olson M, Cooper C. Excess mortality following hip fracture: a systematic epidemiological review. Osteoporos Int. 2009 Oct;20(10):1633-50. doi: 10.1007/s00198-009-0920-3. Epub 2009 May 7. PMID 19421703
- [Background] Kanis JA, Oden A, Johansson H, Borgstrom F, Strom O, McCloskey E. FRAX and its applications to clinical practice. Bone. 2009 May;44(5):734-43. doi: 10.1016/j.bone.2009.01.373. Epub 2009 Feb 3. PMID 19195497
- See also: Company website — http://www.agnovos.com